CLINICAL TRIAL: NCT04696939
Title: Clinical Study of Programmed Cell Death Ligand-1(PD-L1) Antibody (Atezolizumab) Plus Chemotherapy (Carboplatin Plus Etoposide) for Previously Untreated Small Cell Lung Cancer
Brief Title: Combined Atezolizumab and Chemotherapy (Carboplatin Plus Etoposide) in Neoadjuvant Treating Limited-Stage Small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020LY032
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Small-cell Lung Cancer; Neoadjuvant Therapy
Keywords: Limited-Stage Small Cell Lung Cancer; Atezolizumab; Immunotherapy; Carboplatin; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Carboplatin +Etoposide +surgery (Experimental): Neoadjuvant therapy: Atezolizumab, 1200 milligrams(mg) on Day 1 of every 21-day cycle, 2 cycles; Carboplatin, 75 mg per square meter(mg/m^2) on Day 1 of every 21-day cycle, 2 cycles; Etoposide, 100 mg/m^2 on Day 1 of every 3-day cycle, 2 cycles.
  Surgery: patients will receive surgery.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Carboplatin +Etoposide +surgery (Active Comparator): Neoadjuvant therapy: Carboplatin, 75 mg/m^2 on Day 1 of every 21-day cycle, 2 cycles; Etoposide, 100 mg/m^2 on Day 1 of every 3-day cycle, 2 cycles.
  Surgery: patients will receive surgery.
  Interventions: Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab intravenous infusion was administered at a dose of 1200mg on Day 1 of each 21-day cycle.
  Arms: Atezolizumab + Carboplatin +Etoposide +surgery
Drug: Carboplatin — Carboplatin intravenous infusion was administered at a dose of 75mg/m^2 on Day 1 of each 21-day cycle.
Drug: Etoposide — Etoposide intravenous infusion was administered at a dose of 100 mg/m^2 on Day 1 of every 3-day cycle.

SUMMARY:
This Phase II study was designed to evaluate the safety and efficacy of Atezolizumab in combination with Chemotherapy compared with treatment with Chemotherapy alone in previously untreated Limited-Stage Small Cell Lung Cancer patients.

DETAILED DESCRIPTION:
This Phase II study was designed to evaluate the safety and efficacy of Atezolizumab in combination with Chemotherapy (Carboplatin plus Etoposide) compared with treatment with Chemotherapy (Carboplatin plus Etoposide) alone in previously untreated Limited-Stage Small Cell Lung Cancer patients. Participants will be divided in a 1:1 ratio to receive either Atezolizumab + Carboplatin + Etoposide or Carboplatin + Etoposide followed by radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be volunteered to participate in the clinical trial. Patients must sign the informed Consent form (ICF) and be willing to follow and able to complete all test procedures.
2. Histologically or cytologically confirmed stage IIb-IIIb SCLC.
3. Patients with good physical condition and good organ function.
4. Previously untreated patients.
5. Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
6. Patients can tolerate chemotherapy, immunotherapy, and surgery.

Exclusion Criteria:

1. Unclear diagnosis of SCLC.
2. Contraindicated chemotherapy, immunotherapy, and surgery.
3. Undergoing other active malignancies within 5 years or at the same time.Patients with localized curable tumors, such as basal cell carcinoma, squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, or breast carcinoma in situ, will not be excluded.
4. Positive test result for human immunodeficiency virus (HIV).
5. Positive test result for active tuberculosis.
6. Pregnant or lactating women
7. A history of psychotropic substance abuse, drug abuse, or alcoholism.
8. Other factors assessed by the sponsors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival（DFS） | 12 months
  To assess disease free survival（DFS）after surgery.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 3 months
  To assess disease control rate (DCR) after treatment.
Overall survival (OS) | 24 months
  To estimate overall survival (OS) of patients with ES-SCLC.
Objective response rate (ORR) | 3 months
  To evaluate objective response rate (ORR)after treatment.
Duration of response (DOR) | 3 months
  To evaluate duration of response (DOR) after treatment.
Major pathological response (MPR) | 3 months
  To evaluate major pathological response (MPR) after treatment.
Complete pathological response (CPR） | 3 months
  To evaluate complete pathological response (CPR）after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Doctor, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Yang CJ, Chan DY, Shah SA, Yerokun BA, Wang XF, D'Amico TA, Berry MF, Harpole DH Jr. Long-term Survival After Surgery Compared With Concurrent Chemoradiation for Node-negative Small Cell Lung Cancer. Ann Surg. 2018 Dec;268(6):1105-1112. doi: 10.1097/SLA.0000000000002287. PMID 28475559
- [Background] Yang CJ, Chan DY, Speicher PJ, Gulack BC, Tong BC, Hartwig MG, Kelsey CR, D'Amico TA, Berry MF, Harpole DH. Surgery Versus Optimal Medical Management for N1 Small Cell Lung Cancer. Ann Thorac Surg. 2017 Jun;103(6):1767-1772. doi: 10.1016/j.athoracsur.2017.01.043. Epub 2017 Apr 25. PMID 28385378
- [Background] Faivre-Finn C, Snee M, Ashcroft L, Appel W, Barlesi F, Bhatnagar A, Bezjak A, Cardenal F, Fournel P, Harden S, Le Pechoux C, McMenemin R, Mohammed N, O'Brien M, Pantarotto J, Surmont V, Van Meerbeeck JP, Woll PJ, Lorigan P, Blackhall F; CONVERT Study Team. Concurrent once-daily versus twice-daily chemoradiotherapy in patients with limited-stage small-cell lung cancer (CONVERT): an open-label, phase 3, randomised, superiority trial. Lancet Oncol. 2017 Aug;18(8):1116-1125. doi: 10.1016/S1470-2045(17)30318-2. Epub 2017 Jun 20. PMID 28642008